CLINICAL TRIAL: NCT00001747
Title: Racial Differences in Flow Mediated Vasodilator Function
Brief Title: Racial Differences in Control of Blood Vessel Tone and Blood Flow
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980112; 98-H-0112
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Atherosclerosis; Healthy; Hypertension
Keywords: Brachial Artery; Doppler; Endothelium; Nitric Oxide; Nitroglycerin; Normal Volunteer
MeSH Terms: conditions — Atherosclerosis; Hypertension

SUMMARY:
Black Americans tend to die more often from and have more diseases associated with heart disease than White Americans. The exact cause of this is unknown, but it is likely a combination of genetics, behavior, risk factors, strategies for education and prevention, and socioeconomic factors.

Recent studies have suggested that faster biological processes in blood vessels of Black Americans may be the cause of increased amounts of heart disease. In addition, small blood vessels in Black Americans seem to be less responsive to substances that relax blood vessels, which may explain increased blood pressure levels.

In this study researchers plan to study artery relaxation (dilation) in response substances affecting the cells lining blood vessels (endothelin). Researchers will compare the results of this study in black and white people to find out whether racial differences may contribute to increases in heart disease and heart related deaths in blacks.

DETAILED DESCRIPTION:
Black Americans have a greater morbidity and mortality related to cardiovascular diseases compared to whites. The cause for this phenomenon is probably multifactorial and includes differences in pathogenesis, risk factor patterns, genetic background, behavioral variables, strategies for education and prevention, and socioeconomic factors. Recent evidence suggests that acceleration of some of the processes related to vascular biology may account for the greater prevalence of cardiovascular disease in blacks. A diminished vasodilator response of the microvasculature has been shown in African Americans and may therefore be responsible for their increased prevalence of hypertension. Endothelial dysfunction is a central mechanism in the development of atherosclerosis. It is therefore reasonable to postulate that endothelial dysfunction of large conductance arteries may also contribute to a greater susceptibility to atherosclerosis in blacks compared to whites, even in those individuals without the known risk factors for coronary heart disease. In the present study, we propose to investigate brachial artery dilation in response to endothelium-dependent and -independent stimuli in black and white individuals to determine whether racial differences in the vascular biology of large conductance vessels that might contribute to the greater cardiovascular morbidity and mortality previously reported in blacks.

ELIGIBILITY:
Black and white normal volunteers, approximately matched for age and sex, will be included in the study.

All subjects must be capable of rendering informed consent for all procedures.

Volunteers with a history or evidence of present or past hypertension (BP greater than 140/90), diabetes mellitus, hypercholesterolemia (plasma cholesterol greater than 200 mg/dL), cardiac disease, peripheral vascular disease, coagulopathy, chronic smoking (2 pack-years or more), obesity (20% greater than ideal body weight), hyperhomocysteinemia (plasma homocysteine greater than 17 umol/1) or any other disease predisposing them to vasculitis will be excluded from the study.

No pregnant women.

Volunteers who are taking any medication will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108
Dates: Start 1998-05; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hutchinson RG, Watson RL, Davis CE, Barnes R, Brown S, Romm F, Spencer JM, Tyroler HA, Wu K. Racial differences in risk factors for atherosclerosis. The ARIC Study. Atherosclerosis Risk in Communities. Angiology. 1997 Apr;48(4):279-90. doi: 10.1177/000331979704800401. PMID 9112876
- [Background] Geronimus AT, Bound J, Waidmann TA, Hillemeier MM, Burns PB. Excess mortality among blacks and whites in the United States. N Engl J Med. 1996 Nov 21;335(21):1552-8. doi: 10.1056/NEJM199611213352102. PMID 8900087
- [Background] Fang J, Madhavan S, Alderman MH. The association between birthplace and mortality from cardiovascular causes among black and white residents of New York City. N Engl J Med. 1996 Nov 21;335(21):1545-51. doi: 10.1056/NEJM199611213352101. PMID 8900086
- [Derived] Tsimikas S, Szarek M, Cobbaert CM, Romijn F, Jukema JW, Bhatt DL, Bittner VA, Diaz R, Fazio S, Garon G, Yuan C, Gong XM, Goodman SG, White HD, Witztum JL, Steg PG, Schwartz GG; ODYSSEY OUTCOMES Investigators. Oxidized Phospholipids, Lipoprotein(a), and Cardiovascular Outcomes After Acute Coronary Syndrome. Circulation. 2025 Dec 16;152(24):1666-1678. doi: 10.1161/CIRCULATIONAHA.125.073855. Epub 2025 Dec 1. PMID 41321238
- [Derived] van Ommen AM, Diez Benavente E, Onland-Moret NC, Valstar GB, Cramer MJ, Rutten FH, Teske AJ, Menken R, Hofstra L, Tulevski II, Sweitzer N, Somsen GA, den Ruijter HM. Plasma Proteomic Patterns Show Sex Differences in Early Concentric Left Ventricular Remodeling. Circ Heart Fail. 2023 Jul;16(7):e010255. doi: 10.1161/CIRCHEARTFAILURE.122.010255. Epub 2023 Jun 29. PMID 37381923
- [Derived] Maruyama M, Yamamoto T, Abe J, Yodogawa K, Seino Y, Atarashi H, Shimizu W. Number needed to entrain: a new criterion for entrainment mapping in patients with intra-atrial reentrant tachycardia. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):490-6. doi: 10.1161/CIRCEP.113.001416. Epub 2014 Apr 24. PMID 24762806